CLINICAL TRIAL: NCT02176005
Title: Influence of the Administration of DAV132 7.5g Tid for 7 Days on the Fecal Levels of Moxifloxacin During and After a 5-day Oral Treatment With Moxifloxacin 400mg Oad in Healthy Volunteers
Brief Title: Safety and Efficacy Study of DAV132 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Da Volterra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAV132-CL-1002; ID-RCB number 2013-A01504-41 (Other: ANSM (French Agency))
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Moxifloxacin (Active Comparator): Moxifloxacin, oral tablets, 400mg/day, once daily 5 days
  Interventions: Drug: Moxifloxacin
- moxifloxacin + DAV132 (Experimental): Moxifloxacin : 400mg/day for 5 days DAV132: 7.5g x3/day for 7 days
  Interventions: Device: DAV132; Drug: Moxifloxacin
- DAV132 (Experimental): DAV132 oral, 7.5g x3/day for 7 days
  Interventions: Device: DAV132
- Negative control (Placebo Comparator): Negative control: 7.5g x3/day for 7 days
  Interventions: Other: Negative Control

INTERVENTIONS:
Device: DAV132 — DAV132 is associated to moxifloxacin or it is evaluated alone
  Arms: DAV132; moxifloxacin + DAV132
Drug: Moxifloxacin — Moxifloxacin is used alone or associated to DAV132
  Other Names: Avelox
  Arms: Moxifloxacin; moxifloxacin + DAV132
Other: Negative Control — Moxifloxacin is used alone
  Arms: Negative control

SUMMARY:
The purpose of this study is to determine whether DAV132 is safe and effective for capturing fecal residues of moxifloxacin in healthy volunteers.

DETAILED DESCRIPTION:
The proposed study, DAV132-CL-1002, is to evaluate performances of DAV132 in healthy volunteers:

* To capture residual concentration of antibiotics in colon without interfering with their systemic pharmacokinetics parameters.
* To explore the influence of DAV132 to prevent the modification of gut flora due to antibiotic.

In addition, the security and acceptability of DAV132 used during 7 days will be evaluated.

The proposed study is prospective, randomized, controlled, four parallel groups, repeated doses, open-label study blinded to analytical and microbiological evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Normal digestive transit, with usually one daily stool.
* Females participating in the study :

must be either of non-child bearing potential (surgically sterilized at least 3 months prior to inclusion, or postmenopausal or having a negative pregnancy test and be not breastfeeding at screening, and using abstinence or a double contraception method during the treatment period and for additional period of 2 weeks after the end of investigational treatment.

* Having given and signed the written study informed consent prior to undertaking any study-related procedure.
* Covered by the French Health Insurance system.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, haematological, neurological, bone and joint, muscular, psychiatric, systemic, ocular, gynaecologic (if female), or infectious disease, or signs of acute illness.
* Contra-indications to fluoroquinolones, or risk factors for adverse events associated to fluoroquinolones.
* Subjects with a family history of, or actual glucose-6-phosphate dehydrogenase deficiency should be excluded.
* Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should be excluded.
* Contra-indications to DAV132, risk of gastrointestinal obstruction, perforation or haemorrhage, recent digestive tract surgery.
* Fecal colonisation by Clostridium difficile.
* Recent history of hospitalisation (within 3 months prior to inclusion).
* Any antibiotic administration within 3 months before inclusion.
* Any vaccination within the last 28 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Duval, MD, Principal Investigator — CIC Bichat, Paris France
Locations (1):
- CLINICAL INVESTIGATION CENTER (CIC), Groupe Hospitalier Bichat-Claude Bernard, Paris, France

REFERENCES:
- [Background] Edlund C, Beyer G, Hiemer-Bau M, Ziege S, Lode H, Nord CE. Comparative effects of moxifloxacin and clarithromycin on the normal intestinal microflora. Scand J Infect Dis. 2000;32(1):81-5. doi: 10.1080/00365540050164272. PMID 10716083
- [Background] Burkhardt O, Borner K, Stass H, Beyer G, Allewelt M, Nord CE, Lode H. Single- and multiple-dose pharmacokinetics of oral moxifloxacin and clarithromycin, and concentrations in serum, saliva and faeces. Scand J Infect Dis. 2002;34(12):898-903. doi: 10.1080/0036554021000026963. PMID 12587622
- [Derived] de Gunzburg J, Ghozlane A, Ducher A, Le Chatelier E, Duval X, Ruppe E, Armand-Lefevre L, Sablier-Gallis F, Burdet C, Alavoine L, Chachaty E, Augustin V, Varastet M, Levenez F, Kennedy S, Pons N, Mentre F, Andremont A. Protection of the Human Gut Microbiome From Antibiotics. J Infect Dis. 2018 Jan 30;217(4):628-636. doi: 10.1093/infdis/jix604. PMID 29186529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited from March 20th, 2014 (date of first enrolment) and October 17th, 2014 (date of last completed)
Groups:
- Moxifloxacin: Moxifloxacin (oral tablets, 400mg x1/day for 5 days) used alone
- DAV132 + Moxifloxacin: DAV132 (7.5g x3/day taken orally for 7 days) associated to Moxifloxacin (400mg x1/day taken orally for 5 days)
- DAV132: DAV132 (7.5g x3/day taken orally for 7 days) used alone
- Negative Control: Negative control: microcrystalline cellulose (7.5g x3/day taken orally for 7 days)
Period: Overall Study
Arm/Group | Moxifloxacin | DAV132 + Moxifloxacin | DAV132 | Negative Control
Started | 14 | 14 | 8 | 8
Completed | 14 | 14 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moxifloxacin: Moxifloxacin (400mg x1/day taken orally for 5 days) used alone
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin | DAV132 + Moxifloxacin | DAV132 | Negative Control | Total
Number analyzed (Participants) | 14 | 14 | 8 | 8 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (10.4) | 38.6 (12.1) | 27.9 (9.1) | 36.7 (11.8) | 35.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 4 | 5 | 28
  Male | 5 | 4 | 4 | 3 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  France | 14 | 14 | 8 | 8 | 44
Body Mass Index (BMI) at screening visit [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (3.3) | 24.9 (3.2) | 23.6 (3.2) | 23.3 (2.0) | 24.1 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Moxifloxacin Fecal Pharmacokinetics: Area Under the Free Moxifloxacin Fecal Concentration-time Curve Over the Period Time From Beginning of Treatment to 16 Days After the Beginning of Treatment (AUC D1-D16)
Time Frame: D1 pre-dose, D2, D3, D4, D5, D6, D7, D8, D9, D12, D16
Measure: Mean (Standard Deviation); unit: μg/g.day
Arm/Group | Moxifloxacin | Moxifloxacin + DAV132
Number analyzed (Participants) | 14 | 14
μg/g.day | 758.4 (359.3) | 8.28 (7.21)
Statistical Analysis 1: Comparison: Moxifloxacin vs Moxifloxacin + DAV132; Test type: Other; p < .000001, General linear model; Contrast (B/A) = 0.0093, 95% CI 2-sided [0.0060 to 0.0144]

2. Secondary Outcome: Moxifloxacin Fecal Pharmacokinetics: Area Under the Free Moxifloxacin Fecal Concentration-time Curve Over the Period Time From Beginning of Treatment to 37 Days After the Beginning of Treatment (AUC D1-D37)
Time Frame: D1 pre-dose, D2, D3, D4, D5, D6, D7, D8, D9, D12, D16, D23, D30, D37
Measure: Mean (Standard Deviation); unit: μg/g.day
Arm/Group | Moxifloxacin | Moxifloxacin + DAV132
Number analyzed (Participants) | 14 | 14
μg/g.day | 758.7 (359.5) | 8.74 (7.73)
Statistical Analysis 1: Comparison: Moxifloxacin vs Moxifloxacin + DAV132; Test type: Other; p < .000001, General linear model; Contrast (B/A) = 0.0096, 95% CI 2-sided [0.0061 to 0.0151]

3. Secondary Outcome: Moxifloxacin Plasma Pharmacokinetics: AUC(0-24h) of Moxifloxacin Plasma Concentrations Over Time on D1
Time Frame: D1: at pre-dose; 0h30; 1h; 1h30; 2h; 3h; 4h; 6h; 12h and 24h post-dose
Measure: Mean (Standard Deviation); unit: µg/mL.h
Arm/Group | Moxifloxacin | Moxifloxacin + DAV132
Number analyzed (Participants) | 14 | 14
µg/mL.h | 42.1 (7.01) | 41.9 (9.57)
Statistical Analysis 1: Comparison: Moxifloxacin vs Moxifloxacin + DAV132; Test type: Other; p = 0.806, General linear model; Contrast (B/A) = 0.9811, 95% CI 2-sided [0.8608 to 1.1182]

4. Secondary Outcome: Moxifloxacin Plasma Pharmacokinetics: AUC(0-24h) of Moxifloxacin Plasma Concentrations Over Time on D5
Time Frame: D5: at pre-dose; 0h30; 1h; 1h30; 2h; 3h; 4h; 6h; 12h; 24h; 32h; 48h; 56h and 72h post-dose
Measure: Mean (Standard Deviation); unit: µg/mL.h
Arm/Group | Moxifloxacin | Moxifloxacin + DAV132
Number analyzed (Participants) | 14 | 14
µg/mL.h | 57.6 (13.83) | 50.5 (10.91)
Statistical Analysis 1: Comparison: Moxifloxacin vs Moxifloxacin + DAV132; Test type: Other; p = 0.139, General linear model; Contrast (B/A) = 0.8785, 95% CI 2-sided [0.7600 to 1.0155]

5. Secondary Outcome: Moxifloxacin Plasma Pharmacokinetics: Cmax of Moxifloxacin in Plasma on D1
Time Frame: D1: at pre-dose; 0h30; 1h; 1h30; 2h; 3h; 4h; 6h; 12h and 24h post-dose
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Moxifloxacin | Moxifloxacin + DAV132
Number analyzed (Participants) | 14 | 14
µg/mL | 4.02 (1.33) | 4.63 (0.97)
Statistical Analysis 1: Comparison: Moxifloxacin vs Moxifloxacin + DAV132; Test type: Other; p = 0.104, General linear model; Contrast (B/A) = 1.1763, 95% CI 2-sided [0.9982 to 1.3861]

6. Secondary Outcome: Moxifloxacin Plasma Pharmacokinetics: Cmax of Moxifloxacin in Plasma on D5
Time Frame: D5: at pre-dose; 0h30; 1h; 1h30; 2h; 3h; 4h; 6h; 12h; 24h; 32h; 48h; 56h and 72h post-dose
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Moxifloxacin | Moxifloxacin + DAV132
Number analyzed (Participants) | 14 | 14
µg/mL | 4.89 (1.21) | 4.60 (1.24)
Statistical Analysis 1: Comparison: Moxifloxacin vs Moxifloxacin + DAV132; Test type: Other; p = 0.519, General linear model; Contrast (B/A) = 0.9391, 95% CI 2-sided [0.7969 to 1.1066]

7. Secondary Outcome: Number of Adverse Events (Including Abnormal Laboratory Findings) Related to Study Product
Time Frame: From randomization to 37 days after the beginning of treatment
Measure: Number; unit: events related to study product
Arm/Group | Moxifloxacin | Moxifloxacin + DAV132 | DAV132 | Negative Control
Number analyzed (Participants) | 14 | 14 | 8 | 8
events related to study product | 1 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Subjects With Adverse Events Related to Study Product
Time Frame: From randomization to 37 days after the beginning of treatment
Measure: Number; unit: % of subjects with at last 1 related AE
Arm/Group | Moxifloxacin | Moxifloxacin + DAV132 | DAV132 | Negative Control
Number analyzed (Participants) | 14 | 14 | 8 | 8
% of subjects with at last 1 related AE | 7.14 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment period: - 5 days for Moxifloxacin group; - 7 days for the 3 other groups (DAV132 + Moxifloxacin, DAV132 and Negative Control groups)
Groups:
- Moxifloxacin + DAV132: DAV132 (7.5g x3/day taken orally for 7 days) associated to Moxifloxacin (400mg x1/day taken orally for 5 days)
Arm/Group | Moxifloxacin | Moxifloxacin + DAV132 | DAV132 | Negative Control
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/14 | 10/14 | 2/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moxifloxacin (N=14) | Moxifloxacin + DAV132 (N=14) | DAV132 (N=8) | Negative Control (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intestinal transit time abnormal (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Formication (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less